CLINICAL TRIAL: NCT07108972
Title: Comparison Between Laparoscopic Transabdominal Pre-peritoneal (TAPP) Versus Total Extraperitoneal (TEP) for Inguinal Hernia Repair.
Brief Title: Laparoscopic Inguinal Hernia Repair TEP vs TAPP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Moamen Hassan Ezeldin, Principal Investigator, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-2-04MS
Record Dates: First submitted 2025-07-23; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Laparoscopic Inguinal Hernia Repair

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAPP Group (Active Comparator)
  Interventions: Procedure: Transabdominal pre-peritoneal laparoscopic inguinal hernia repair
- TEP Group (Active Comparator)
  Interventions: Procedure: Totally extraperitoneal laparoscopic inguinal hernia repair

INTERVENTIONS:
Procedure: Transabdominal pre-peritoneal laparoscopic inguinal hernia repair — laparoscopic inguinal hernia repair surgical technique that it's main principal is placing the mesh pre-peritoneally through transabdominal approach
  Arms: TAPP Group
Procedure: Totally extraperitoneal laparoscopic inguinal hernia repair — laparoscopic inguinal hernia repair surgical technique that it's main principal is placing the mesh pre-peritoneally through extraperitoneal approach
  Arms: TEP Group

SUMMARY:
This study is dedicated to compare between 2 different techniques is the management of inguinal hernia repair using laparoscopic intervention and how it may affect the patients life style covering both benefits and possible adverse affects for each method

ELIGIBILITY:
Inclusion Criteria

- All patients with inguinal hernias (direct and indirect ؛pubonocele type/funicular type؛) with age between 15 to 60 years and any sex at the period between May 2024 to May 2025 presented electively to the outpatient clinic of the department of General surgery, Sohag University Hospital

Exclusion Criteria:

* Patients with age below 15 years and more than 60 years.
* Patients with mega hernias or complete indirect inguinal hernia.
* Patients with obstructed or strangulated inguinal hernia.
* Patients with abdominal malignancy & cirrhosis with end stage liver disease.
* Pregnancy or planning to become pregnant.
* History of forced hernial reduction.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Persisting pain | post-operatively up to 8 weeks
  a specific questionnaire will be used to assess the extent and nature of pain post-operative
Hernia recurrence | post-operatively up to 6 months

SECONDARY OUTCOMES:
Duration of operation (min) | Baseline
Length of hospital stay (Days) | up to 2 weeks
Time to return to usual activities (Days) | Post-operatively up to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No